CLINICAL TRIAL: NCT00602433
Title: Evaluation of Hormonal Changes in Women on Erlotinib Therapy
Brief Title: Hormone Changes in Women With Stage IIIB or Stage IV Non-Small Cell Lung Cancer Receiving Erlotinib
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Jyoti Patel, MD, Northwestern University
Other Study IDs: NU 07CC4; STU00001887 (Other: Northwestern University IRB)
Record Dates: First submitted 2008-01-17; First posted 2008-01-28 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Advanced Nonsmall Cell Lung Cancer
Keywords: advanced nonsmall cell lung cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood will be tested for different sex hormones as well as glucose metabolism
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- questionnaire and laboratory biomarker analysis: Subjects with advanced non-small cell lung cancer and take erlotinib as part of their anticancer therapy for at least 3 months. Subjects have had some changes in hair growth, acne or menses (periods) that might be a side effect of erlotinib. Subjects will complete a questionnaire and blood collected for biomarker analysis.

SUMMARY:
Studying samples of blood in the laboratory from patients receiving erlotinib may help doctors learn more about the effects of erlotinib on hormone levels.

This clinical trial is looking at hormone changes in women with stage IIIB or stage IV non-small cell lung cancer receiving erlotinib.

DETAILED DESCRIPTION:
Patients undergo a dermatology evaluation and complete the Polycystic Ovarian Syndrome (PCOS) research study questionnaire once. Blood samples are collected after an overnight fast. Samples are analyzed for circulating levels of total and bioavailable testosterone, dehydroepiandrosterone sulfate, and sex hormone binding globulin. Serum luteinizing hormone, follicle stimulating hormone, fasting glucose, and insulin levels are also assessed.

ELIGIBILITY:
* Histologically confirmed non-small cell lung cancer

  * Stage IIIB (effusion) or stage IV disease
* Must be receiving daily erlotinib hydrochloride for more than 3 months
* Must have hirsutism, acne, androgenic alopecia, amenorrhea, truncal weight gain, or other clinical phenotype associated with syndrome of androgen excess

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects have advanced nonsmall cell lung cancer and have been taking erlotinib as part of anticancer therapy for at least 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2007-12; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Presence of hyperandrogenemia | One approximate 30 minute visit
  We will determine if hyperandrogenemia is present in women with nonsmall cell lung cancer who are taking erlotinib.

SECONDARY OUTCOMES:
Dermatologic manifestations | One approximate 30 minute visit
  We will describe the dermatologic manifestations of erlotinib in women
Changes in body habitus and patterns of hair loss | One approximate 30 minute visit
  We will describe changes in body habitus and patterns of hair loss from women on erlotinib.

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti D. Patel, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Northwestern Medical Faculty Foundation, Chicago, Illinois, United States